CLINICAL TRIAL: NCT04291053
Title: The Efficacy and Safety of Huai er in the Adjuvant Treatment of COVID-19: a Prospective, Multicenter, Randomized, Parallel Controlled Clinical Study
Brief Title: The Efficacy and Safety of Huai er in the Adjuvant Treatment of COVID-19
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Chen Xiaoping, Principal Investigator, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJ-IRB20200205
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: COVID-19
Keywords: COVID-19; Huaier granule
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Standard therapy+Huaier granule Huaier granule 20g, po, tid for 2 weeks( or until discharge)
  Interventions: Drug: Huaier Granule
- control group (No Intervention): standard therapy

INTERVENTIONS:
Drug: Huaier Granule — standard treatment + Huaier Granule 20g po tid for 2weeks
  Arms: experimental group

SUMMARY:
In December 2019,a new type of pneumonia caused by the coronavirus (COVID-2019) broke out in Wuhan ,China, and spreads quickly to other Chinese cities and 28 countries. More than 70000 people were infected and over 2000 people died all over the world.There is no specific drug treatment for this disease. This study is planned to observe the efficacy and safety of Huaier granule in the adjuvant treatment COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 75 years, extremes included, male or female
2. Patients diagnosed with mild or common type COVID-19, according to the official guideline "Pneumonia Diagnosis and Treatment Scheme for Novel Coronavirus Infection (Trial Version 6)"
3. patients can generally tolerable for treatment recommended by the official guideline "Pneumonia Diagnosis and Treatment Scheme for Novel Coronavirus Infection (Trial Version 6)"
4. Patients have not been accompanied by serious physical diseases of heart, lung, brain, etc.,Eastern Cooperative Oncology Group score standard:0-1
5. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Female subjects who are pregnant or breastfeeding.
2. patients who are allergic to this medicine
3. patients meet the contraindications of Huaier granule
4. Patients with diabetes
5. Patients have any condition that in the judgement of the Investigators would make the subject inappropriate for entry into this study.
6. patients can't take drugs orally

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Mortality rate | up to 28 days
  All cause mortality

SECONDARY OUTCOMES:
Clinical status assessed according to the official guideline | up to 28 days
  1.mild type：no No symptoms, Imaging examination showed no signs of pneumonia; 2,moderate type: with fever or respiratory symptoms,Imaging examination showed signs of pneumonia, SpO2>93% without oxygen inhalation ; severe type:Match any of the following：a. R≥30bpm；b.Pulse Oxygen Saturation(SpO2)≤93% without oxygen inhalation，c. PaO2/FiO2(fraction of inspired oxygen )≤300mmHg ；4. Critically type：match any of the follow: a. need mechanical ventilation; b. shock; c. (multiple organ dysfunction syndrome) MODS
The differences in oxygen intake methods | up to 28 days
  Pulse Oxygen Saturation(SpO2)>93%，1. No need for supplemental oxygenation; 2. nasal catheter oxygen inhalation（oxygen concentration%,The oxygen flow rate：L/min）；3. Mask oxygen inhalation（oxygen concentration%,The oxygen flow rate：L/min）；4. Noninvasive ventilator oxygen supply（Ventilation mode,oxygen concentration%,The oxygen flow rate：L/min,）；5. Invasive ventilator oxygen supply（Ventilation mode,oxygen concentration%,The oxygen flow rate：L/min,）.
Duration (days) of supplemental oxygenation | up to 28 days
  days
Duration (days) of mechanical ventilation | up to 28 days
  days
The mean PaO2/FiO2 | up to 28 days
Length of hospital stay (days) | up to 28 days
  days
Length of ICU stay (days) | up to 28 days
  days
Pulmonary function | up to 3 months after discharge
  forced expiratory volume at one second ,maximum voluntary ventilation at 1month，2month，3month after discharge